CLINICAL TRIAL: NCT02130167
Title: Low Concentrations of Atropine for Controlling Myopia Progression in School Children
Brief Title: Low Concentration Atropine for Myopia Progression in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8C0601
Record Dates: First submitted 2014-04-28; First posted 2014-05-05 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Myopia Progression
Keywords: Myopia progression; Low concentration atropine
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.01% Atropine (Experimental)
  Interventions: Drug: Atropine
- 0.05% Atropine (Active Comparator)
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Compare different concentrations of atropine eye drops (0.01% vs 0.05%) in the efficacy of controlling myopia progression and side effects of atropine

SUMMARY:
Myopia is the leading cause of blindness in Taiwan. The younger children with myopia, the higher risk of high myopia in later life and complications such as retinal detachment and maculopathy will occur. We have reported the low concentration of atropine (0.05%) with the effect on retarding the myopia progression. Recently the 0.01% atropine was also reported effective and with less visual side effects such as mydriasis. The aim of this study is to compare the efficacy in controlling myopia progression and visual side effects of 2 low concentration of atropine(0.05% vs 0.01%) in children aged 6-12 years with myopia of at least -0.5 diopters (D) and astigmatism of -1.50 D or less.

ELIGIBILITY:
Inclusion Criteria:

Myopia of at least -0.5 diopters (D) and astigmatism of -1.50 D or less.

Exclusion Criteria:

strabismus, amblyopia. cataract, glaucoma or any ocular diseases ocular surgery history systemic diseases (ex. asthma, heart disease...)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cycloplegic spherical refraction change | 1 year
  Cycloplegic spherical refraction change is the main indicator of the myopia progression.

SECONDARY OUTCOMES:
Axial length change | 1 year
  Axial length change is another indicator of the myopia progression.Using non-contact biometry. unit: millimeter(mm)

OTHER OUTCOMES:
pupil size | 6 months
  Using computer scaling software. unit: millimeter(mm)
accommodation | 6 months
  Using accommodometer to measuer accommodation. Unit: diopeter
Questionnaire | baseline and 6 months
  Questionnaire written by patients and their parents about how many hours per week of near work (ex. computer/video game, reading, piano playing...) and outdoor activities, the compliance of atropine use, discomfort after atropine use (ex. photophobia or blurred vision when near work)

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Chang Wu, MD,PhD, Principal Investigator — Dep. of Ophthalmology, Kaohsiung Chang Gung Memorial Hospital, Taiwan
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan